CLINICAL TRIAL: NCT05816759
Title: A Randomized, Open-label, Single Oral Dosing, Two-sequence, and Two-period Crossover Study to Evaluate the Pharmacokinetics and Safety Between the Administration of CKD-383 and the Co-administration of CKD-501, D744, and D150 for Healthy Subjects in Fed State
Brief Title: Evaluate the Pharmacokinetics and Safety Between the Administration of CKD-383 and the Co-administration of CKD-501, D744, and D150
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A101_04BE2113
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: CKD-383 (A single oral dose of 1 tablet under fed condition) Period 2: CKD-501, D744, D150 (A single oral dose of 3 tablets under fed condition)
  Interventions: Drug: CKD-383; Drug: CKD-501, D744, D150
- Sequence B (Experimental): Period 1: CKD-501, D744, D150 (A single oral dose of 3 tablets under fed condition) Period 2: CKD-383 (A single oral dose of 1 tablet under fed condition)
  Interventions: Drug: CKD-383; Drug: CKD-501, D744, D150

INTERVENTIONS:
Drug: CKD-383 — QD, PO
Drug: CKD-501, D744, D150 — QD, PO

SUMMARY:
Evaluate the Pharmacokinetics and Safety Between the Administration of CKD-383 and the Co-administration of CKD-501, D744, and D150 for Healthy Subjects in Fed State

ELIGIBILITY:
Inclusion Criteria:

1. Those who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.
2. Healthy adult who aged 19 to 55 years.
3. Those who meet the criteria of anthropometric data

   * Man: Body weight ≥ 50 kg, Body mass index 18 to 30 kg/m2
   * Woman: Body weight ≥ 45 kg, Body mass index 18 to 30 kg/m2

Exclusion Criteria:

1. Those who have medical history of hypersensitivity to active pharmaceutical ingredient (Lobeglitazone, Sitagliptin, Metformin) or additives.
2. Those who have clinically significant disease or medical history of Hepatopathy, Renal dysfunction, Neurological disorder, Immunity disorder, Respiratory disorder, Genitourinary system disorder, Digestive system disorder, Endocrine system disorder, Cardiovascular disorder, Blood tumor, Psychical disorder, Severe urinary tract infection.
3. Those who have past medical history of gastrointestinal disorder (Crohn's disease, ulcerative colitis, etc. except simple appendectomy or hernia surgery), which affect the absorption of drug.
4. Those who have Drug abuse (especially sleeping drugs, central analgesics, opiates or psychotropic drugs such as psychotropic drugs) or persons with a history of substance abuse.
5. Those who have the test results written below

   * AST, ALT > 2 times higher than upper normal level
   * Total bilirubin > 2 times higher than upper normal level
   * eGFR (estimated Glomerular Filtration Rate, which is calculated by MDRD) < 60 mL/min/1.73m2
   * "Positive" or "Reactive" test result of Hepatitis B & C, HIV, RPR
   * Under 5 min resting condition, systolic blood pressure >160 mmHg or <90 mmHg, diastolic blood pressure >100 mmHg or <50 mmHg
6. Those who have determined that the abnormal results are clinically significant in the screening test items (question, vital signs, electrocardiogram, physical test, blood, urine test, etc.).
7. Those who participated in other clinical trials within 180 days of the intended study drug administration and have been administered clinical trial medications (except for those who have not taken the study medication).
8. Those who has taken a drug (Ethical drug, over the counter drug, herbal medicine, or nutritional supplement (vitamin, etc.)) within 14 days prior to screening (however, if it is considered that it does not affect the safety and research results of the subject, as determined by the investigator).
9. Those who donated whole blood within 8 weeks prior to screening, or who donated or donated components (plasma, platelets) within 4 weeks, and consented to prohibit blood donation from 30 days after the last administration of investigational product.
10. Those who have continuously consumed more than 21 units/week (1 unit of alcohol = 10 g = 12.5 mL) within 6 months prior to screening.
11. Those who have More than 10 smokers a day within 6 months prior to screening.
12. Those who cannot use clinically acceptable contraceptive methods (e.g., infertility surgery between themselves and partners, intrauterine contraceptive devices, use of diaphragms or condoms) from the time the drug is administered to the last visit.
13. Those who cannot inhibit the diet (especially grapefruit juice, caffeine) that can affect the absorption, distribution, metabolism, and excretion of the drug from 3 days before the last administration of the investigational product to the last visit.
14. Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
15. Those who receive intravenous administration of radioactive iodine contrast agents (for intravenous urography, venous cholangiography, angiography, computed tomography using contrast agents, etc.) within 48 hours before the first administration of investigational product.
16. Those who are pregnant or breastfeeding.
17. Those who are deemed inappropriate to participate in clinical trial by investigators.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Cmax of CKD-383 | Pre-does(0 hour), Post-dose(0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour)
  Cmax: Maximum plasma concentration of the drug
AUCt of CKD-383 | Pre-does(0 hour), Post-dose(0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour)
  AUCt: Area under the concentration-time curve from time zero to time

CONTACTS AND LOCATIONS:
Overall Officials: Anhye Kim, Ph.D, Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Bundang, South Korea